CLINICAL TRIAL: NCT02508961
Title: WEB-Based Physiotherapy for People With Multiple Sclerosis
Acronym: WEB-PaMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Glasgow (Other)
Collaborators: National Heatlh Service Ayrshire and Arran (Other Government); NHS Lothian (Other Government); University of Plymouth (Other); University Hospital Plymouth NHS Trust (Other)
Responsible Party: Principal Investigator, Dr Lorna Paul, Dr, University of Glasgow
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15/WS/0030
Record Dates: First submitted 2015-07-23; First posted 2015-07-27 (Estimated); Last update posted 2017-06-01 (Actual); Status verified 2017-05

CONDITIONS: Multiple Sclerosis
Keywords: Physical Activity; Exercise; Physiotherapy
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Web-based physio (Experimental): Participants receive an online individualised exercise programme to complete over the internet twice per week. Exercises can be a combination of aerobic, strengthening and balance exercises. Participants receive a weekly phone call from a physiotherapist for the first two weeks to check on progress. After this, every 2 weeks online exercise diaries are remotely monitored by a physiotherapist and exercise programmes progressed as appropriate.
  Interventions: Behavioral: Exercise
- Print-out exercise programme (Active Comparator): Participants receive printed exercise programme to complete twice per week. Exercises can be a combination of aerobic, strengthening and balance exercises. Participants receive a weekly phone call from a physiotherapist for the first two weeks to check on progress. Participants complete a paper exercise diary and after the first 2 weeks if they require a progression to their exercise programme they contact their physiotherapist.
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — web-based physio exercise programme

SUMMARY:
The study will be a pragmatic, single blind, randomised, controlled feasibility study, comparing 6 months of web-based physiotherapy plus usual care with usual care alone in pwMS. The study will recruit 90 pwMS from three UK Centres (30 from each centre); NHS Ayrshire and Arran, NHS Lothian, and Plymouth Hospitals NHS Trust.

The aim of this study is to assess the feasibility of a randomised controlled trial examining the effectiveness of a six-month web-based physiotherapy programme and usual care compared to usual care alone, in people moderately affected by MS and to gather essential information for the planning of a definitive trial, which would evaluate both clinical and cost effectiveness of the intervention.

DETAILED DESCRIPTION:
Following baseline assessments, both groups will be given an appointment with the physiotherapist to agree shared goals and to devise an individualised exercise programme based upon their needs and treatment goals. Participants will then be randomised to one of two groups.

Participants randomised to the intervention group will receive their individualised exercise programme delivered via the web-based physio website. Participants will be asked to complete their exercise programme at least twice weekly. They will receive weekly standardised phone calls from the physiotherapist for the first two weeks of the programme. Every two weeks thereafter for the remainder of the 6 month intervention period the physiotherapist will review the exercise diary of each participant and remotely alter the participant's exercise programme as appropriate, by changing any combination of exercises, level of difficulty or number of repetitions. The number and type of exercises within the programme and duration to complete the exercise programme will be documented. Participants will be informed of any changes by standardised email.

Participants randomised to the control group will receive a print out exercise sheet of their individualised exercise programme. Participants will be asked to complete their exercise programme at least twice weekly. Compliance will be captured using a home exercise diary. Participants will also receive a weekly phone call from the physiotherapist for the first two weeks to check on progress.

ELIGIBILITY:
Inclusion Criteria:

* A confirmed diagnosis of MS
* Known to a MS consultant in NHS Ayrshire and Arran, Lothian or Plymouth Hospitals NHS Trust
* EDSS of 4 - 6.5
* Access to a personal computer/tablet or smart television with an email address and internet connection

Exclusion Criteria:

* Currently taking part in regular exercise (two or more times per week) and/or a regular physiotherapy programme
* Poor cognitive function as assessed by a Mini Mental State Examination Score (MMSE) <24
* Any significant change in medication (within the last 3 months)
* Relapse within 3 months requiring treatment
* Other significant co-morbidities for which exercise is contra-indicated
* Unwilling to be randomised to intervention/control group
* Currently participating in another clinical trial (rehabilitation or pharmacological)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Compliance to the exercise programme | 9 months
  Number of completed exercise diary entries
Two Minute Walk Test | 9 months

SECONDARY OUTCOMES:
Timed 25 Foot Walk | 9 months
Timed Up and Go | 9 months
Berg Balance Scale | 9 months
Physical Activity | 9 months
  Measured using the activPAL physical activity monitor
MS-Related Symptom Checklist | 9 months
Multiple Sclerosis Impact Scale | 9 months
Hospital Anxiety and Depression Scale | 9 months
Health related quality of life | 9 months
  EQ-5D

CONTACTS AND LOCATIONS:
Locations (3):
- United Kingdom (3):
  - Anne Rowling Regenerative Neurology Clinic, Edinburgh
  - Douglas Grant Rehabilitation Centre, Irvine
  - University of Plymouth, Plymouth

REFERENCES:
- [Derived] Dennett R, Coulter E, Paul L, Freeman J. A qualitative exploration of the participants' experience of a web-based physiotherapy program for people with multiple sclerosis: Does it impact on the ability to increase and sustain engagement in physical activity? Disabil Rehabil. 2020 Oct;42(21):3007-3014. doi: 10.1080/09638288.2019.1582717. Epub 2019 Mar 23. PMID 30907159